CLINICAL TRIAL: NCT02997293
Title: An Analysis of the Impact of the Enhanced Recovery After Surgery System for Colorectal Surgery at the University of Arkansas for Medical Sciences
Brief Title: Impact of the Enhanced Recovery After Surgery System for Colorectal Surgery
Status: Recruiting | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 206240
Record Dates: First submitted 2016-12-12; First posted 2016-12-20 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: ColoRectal Cancer and Inflammatory Bowel Disease
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enhanced Recovery: Those subjects who had major colorectal surgery at the University of Arkansas for Medical Sciences after Enhanced Recovery After Surgery implementation, between the dates of June 1, 2015 to November 30, 2016
  Interventions: Other: Enhanced Recovery protocol
- pre-Enhanced Recovery: Those subjects who had major colorectal surgery at the University of Arkansas for Medical Sciences prior to Enhanced Recovery After Surgery implementation between the dates of January 1, 2014 to December 31, 2014
  Interventions: Other: Enhanced Recovery protocol

INTERVENTIONS:
Other: Enhanced Recovery protocol — The Enhanced Recovery protocol focuses on many areas or perioperative care, including non-narcotic pain management, optimization of fluid balance throughout the perioperative course, early eating, ambulation, early removal of drains postoperatively, and preoperative patient education.

SUMMARY:
This is an observational study to look at the impact of the Enhanced Recovery After Surgery system for colorectal surgery (Group 1) in shortening hospital length of stay, reducing postoperative narcotic consumption, lowering Visual Analog Scale scores, decreasing the incidence of postoperative nausea and vomiting, and reducing 30-day readmission when compared to patients who had colorectal surgery performed at UAMS prior to the implementation of the Enhanced Recovery After Surgery system (Group 2).

This is a retrospective study using de-identified records and therefore will not require subject enrollment and is NOT Human Subjects Research.

DETAILED DESCRIPTION:
The Enhanced Recovery After Surgery system for perioperative care of patients undergoing major abdominal surgery, particularly colorectal surgery, was formed in Europe by a surgeon named Henrik Kehlet in 1994. Dr. Kehlet observed that his patients undergoing colorectal surgery were hospitalized postoperatively for extended periods of time due to prolonged return of the normal intestinal physiology and of other bodily functions. Dr. Kehlet formulated a system of perioperative care that focused on preserving and promoting faster return of normal physiologic function of the human body following surgery.

The Enhanced Recovery After Surgery system has been implemented in the United States for nearly a decade now, primarily at major academic institutions. Numerous publications exist that report the dramatic positive impacts of this program on reducing postoperative hospital length of stay, reducing 30-day hospital readmissions, and improving patient satisfaction.

The University of Arkansas for Medical Sciences implemented several components of the Enhanced Recovery After Surgery system for colorectal surgery in June 2015. This is an observational study to look at the impact that program (Group 1) in shortening hospital length of stay, reducing postoperative narcotic consumption, lowering Visual Analog Scale scores, decreasing the incidence of postoperative nausea and vomiting, and reducing 30-day readmission when compared to patients who had colorectal surgery performed at University of Arkansas for Medical Sciences prior to the implementation of the Enhanced Recovery After Surgery system (Group 2).

ELIGIBILITY:
Inclusion Criteria:

* All men and women 18 years and older who underwent major colorectal surgery at University of Arkansas for Medical Sciences between January 1, 2014 to December 31, 2014 and June 1, 2015 to November 30, 2016, and were American Society of Anesthesiologist physical status classification 1-3 at the time of surgery.

Exclusion Criteria:

* American Society of Anesthesiologists physical status classification > 3 and age < 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All men and women 18 years and older who underwent major colorectal surgery at the University of Arkansas for Medical Sciences between January 1, 2014 to December 31, 2014 and June 1, 2015 to November 30, 2016, and were American Society of Anesthesiologist physical status classification 1-3 at the time of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | 30 days from the conclusion of the surgical procedure
  To compare the hospital length of stay following major colorectal surgery at the University of Arkansas for Medical Sciences for patients who had their perioperative care guided by the principles of the Enhanced Recovery After Surgery system to those that had major colorectal surgery at University of Arkansas for Medical Sciences prior to the implementation of the Enhanced Recovery After Surgery system.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Mehaffey, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No